CLINICAL TRIAL: NCT04055246
Title: Measuring Effects of Prebiotics on Human Behavior and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00093322
Record Dates: First submitted 2019-07-26; First posted 2019-08-13 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Prebiotics and Human Behavior and Cognition
MeSH Terms: interventions — Inulin; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (Experimental): Participants receive prebiotics containing fiber bar to consume 2x daily for 1 week.
  Interventions: Dietary Supplement: Inulin
- Placebo (Placebo Comparator): Participants receive placebo bar containing no added prebiotics to consume 2x daily for 1 week.
  Interventions: Dietary Supplement: Placebo (maltodextrin)

INTERVENTIONS:
Dietary Supplement: Inulin — 9 grams of food grade inulin added to custom made fiber bars.
  Arms: Prebiotic
Dietary Supplement: Placebo (maltodextrin) — 9 grams of food grade maltodextrin - replaces inulin in fiber bars.
  Arms: Placebo

SUMMARY:
This study is designed to test the effects of prebiotics on cognition, behavior and physiology in healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of dietary carbohydrate supplements (prebiotics) on cognition, behavior and physiology in healthy individuals.

This study will be separated into one pre-study visit + three consecutive weeks: Baseline (week 1), Intervention (week 2) and Assessment (week 3). For these three weeks, participants will be asked to take diet surveys and make in-person visits to complete online cognitive assessments and provide samples of blood and saliva to assess levels of serotonin and cortisol in addition to other basic metabolites. During the Intervention week, participants will be given snack bars that they will be asked to eat twice a day, for five days in a row. There will be two treatment groups that participants will be randomly assigned to, which vary according to the carbohydrate makeup of snack bars. For the entire three-week study period, participants will also be asked to collect samples of their stool at home every Tuesday and Friday. They will also be provided with wearable devices (a watch) to track their daily heart rate and activity level (including sleep) for the entirety of the study. Participants will be compensated for their time for each stage of the study, once in-person visits begin.

The greatest risks of this study include the possibility of infection while sampling your own stool, and momentary discomfort and/or bruising associated with blood draws. Discomfort as a result of consuming the bars is possible in the form of flatulence, bloating, constipation, diarrhea, or borborygmi (stomach rumbling). Participants weighing less than 140 pounds may be more likely to develop diarrhea than those weighing more. Should any such discomfort occur, it can be alleviated simply by discontinuing consumption of the prebiotic. Infection, fainting, and excess bleeding/clotting, though highly unlikely, are also possible. Participants also face risks associated with the loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18 and 35
* Able to provide stool samples at no risk to yourself
* Weigh at least 110 pounds
* Physically able to perform a cognitive examination administered on a laptop with a trackpad (no significant language, hearing, visual or sensory-motor problems)

Exclusion Criteria:

* History or current diagnosis of acute or active major psychiatric disorder (major depressive disorder, generalized anxiety disorder, post-traumatic stress disorder, schizophrenia, bipolar disorder, alcohol or drug dependence, etc)
* History or current diagnosis of any neurological disorder (convulsion or seizure disorder, epilepsy, Huntington's Disease, Multiple Sclerosis, ALS, Parkinson's, dementia, stroke, etc)
* Use of steroid medications, including but not limited to steroid inhalers or creams or lotions that contain steroids, such as hydrocortisone
* Drink greater than 2 alcoholic beverages per day on average
* Recreational drug use, including but not limited to marijuana, cocaine, ecstasy, etc, within the past month
* Known food allergies to soy products
* Dietary restrictions/allergies of milk or dairy products including food products that do not contain nuts, peanuts, eggs, or shellfish, but was manufactured in the same space as these food allergens
* History or current diagnosis of autism or pervasive development disorder
* History or current diagnosis of any learning disability
* History of fainting during blood draws
* Use chewing tobacco
* Currently pregnant
* Currently breastfeeding
* BMI higher than 27.5 or less than 17
* History or current diagnosis of irritable bowel syndrome
* History or current diagnosis of inflammatory bowel disease
* History or current diagnosis of type 2 diabetes
* History or current diagnosis of chronic kidney disease with decreased kidney function
* History or current diagnosis of intestinal obstruction
* History or current diagnosis of untreated colorectal cancer
* Colonoscopy within the past month
* Oral antibiotics within the past month

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Change in cognitive test performance from baseline | Baseline (Day 2, Day 5), Intervention (Day 9, Day 12), and Post-Intervention (Day 16, Day 19)
  We will measure performance on a ten-domain cognitive battery (score out of 1000 for each domain) and compare the change from baseline between treatment and control groups.
Change in stool microbiota profile from baseline | Baseline (Day 2, Day 5), Intervention (Day 9, Day 12), and Post-Intervention (Day 16, Day 19)
  Stool samples will be analyzed to determine microbiota composition by 16S rRNA sequencing, and we will compare the change from baseline between treatment and control groups.

SECONDARY OUTCOMES:
Change in nighttime salivary cortisol from baseline | Baseline (Day 1, Day 4), Intervention (Day 8, Day 11), and Post-Intervention (Day 15, Day 18)
  Saliva samples will be analyzed for cortisol concentration, and we will compare the change from baseline between treatment and control groups.
Change in blood metabolites from baseline | Baseline (Day 2, Day 5), Intervention (Day 9, Day 12), and Post-Intervention (Day 16, Day 19)
  Blood samples will be analyzed for a panel of metabolites that may be influenced by the intestinal microbiota, and we will compare the change from baseline between treatment and control groups
Change in sleep quality from baseline | Baseline (Days 1-5), Intervention (Days 8-12), and Post-Intervention (Days 15-19)
  Smart watches will be used to monitor time asleep each night and we will compare the change in this variable from baseline between treatment and control groups
Change in sleep quality from baseline | Baseline (Days 1-5), Intervention (Days 8-12), and Post-Intervention (Days 15-19)
  Smart watches will be used to monitor percent of time spent in deep sleepwe will compare the change in this variable from baseline between treatment and control groups
Change in heart rate from baseline | Smart watches will be used to continuously monitor heart rate, and we will compare the change from baseline between treatment and control groups
  Baseline (Days 1-5), Intervention (Days 8-12), and Post-Intervention (Days 15-19)
Change in stool short-chain fatty acid (SCFA) content from baseline | Baseline (Day 2, Day 5), Intervention (Day 9, Day 12), and Post-Intervention (Day 16, Day 19)
  Stool samples will be analyzed to determine initial concentrations of SCFAs and capacity to produce SCFAs in response to a prebiotic intervention in vitro, and we will compare the change from baseline in these variables between treatment and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence David, Ph. D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data at this time.